CLINICAL TRIAL: NCT02251743
Title: Double-Blind 2-Site Randomized Clinical Trial of Neurofeedback for ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of North Carolina (Other)
Responsible Party: Principal Investigator, L. Eugene Arnold, Professor Emeritus of Psychiatry, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013H0417; 1R01MH100144-01A1 (NIH)
Record Dates: First submitted 2014-09-17; First posted 2014-09-29 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: ADHD; Attention-Deficit/Hyperactivity Disorder; neurofeedback; EEG
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neurofeedback treatment (Experimental): The intended treatment is downtraining of theta power and uptraining of beta power for 38 treatments of active NF.
  Interventions: Device: Neurofeedback treatment
- Sham neurofeedback treatment (Placebo Comparator): Participants assigned to sham and their trainers will be fed EEG data from pre-recorded files (recorded during live clinical NF) rather than from the participant's live signal. In order to prevent unblinding of experienced NF trainers/technicians, artifacts from the participant's EMG and EOG are blended into the pre-recorded EEG so that the trainer controlling the feedback cannot differentiate between live and simulated data. To insure trainer/technician blindness, the pre-recorded EEG will be 38 consecutive EEGs from the same age-matched clinical case so that EEGs of the sham group will also show "training progress" over successive sessions, like real NF.
  Interventions: Device: Neurofeedback treatment

INTERVENTIONS:
Device: Neurofeedback treatment — Each session, the child participates in 5 training tasks. Each task lasts 5 minutes at the beginning and gradually increases to 9 minutes per task over the course of the neurofeedback as the child's attention span improves. We record four results for each of the 5 tasks:
  1. The number of half-second periods that they met the reward parameters (i.e. theta mV below threshold; beta mV above threshold)
  2. Average voltage of theta waves
  3. Average voltage of beta
  4. Average ratio of theta to beta power (TBR)

SUMMARY:
Additional treatments with long-term benefit for attention-deficit/hyperactivity disorder (ADHD) are needed; one of the more promising is neurofeedback (EEG biofeedback), which has several randomized controlled trials showing significant benefit, but which are inconclusive because they were not double-blinded; the benefit could have been nonspecific (placebo response). Because of neurofeedback's labor-intensive cost (1 treatment costing as much as a month's medication), It is important to know how much specific benefit it yields. This 2- site placebo-controlled double-blind randomized clinical trial is the first to test for a specific benefit of neurofeedback with adequate power, the first designed and implemented collaboratively by experts in neurofeedback, ADHD, and clinical trials, the first to rigorously monitor quality not only of treatment, but also of placebo and blinding, and the first to follow up for 2 years to examine enduring effect; the results, whether positive or negative, will provide evidence for clinical practice and public policy regarding ADHD.

DETAILED DESCRIPTION:
Current established, evidence-based treatments for attention-deficit/hyperactivity disorder (ADHD) are incompletely effective and not universally acceptable, and appear to wane in effect over time despite significant immediate benefit. E.g., FDA-approved medication, which shows large acute benefit, leaves a third of children only partially treated even when combined with behavioral treatment, and has not been demonstrated effective beyond 2 years. Additional treatments are needed that are effective with persisting benefit, preferably related to a biomarker predicting treatment response. A good candidate is electroencephalographic (EEG) biofeedback, called neurofeedback (NF). It is based on 1) observations that patients with ADHD often have excessive theta band (4-8 Hz) quantitative EEG power, low beta band (13-21 Hz) power, and excessive theta beta ratio (TBR), and 2) theoretical application of operant conditioning to correct this EEG imbalance. Metaanalysis of 6 randomized clinical trials found a large benefit for inattentive symptoms and medium benefit for hyperactive-impulsive symptoms. Unfortunately, none of these were blinded. Three of 4 small blinded studies found no advantage for NF over sham, but used suboptimal NF, leaving the situation inconclusive. Because of the expense and time required by NF, there is a public health need to determine whether it has a specific effect beyond the obvious nonspecific benefit of doing a focused activity several times a week with a friendly,encouraging adult who reinforces for attending to the task. Experts in NF, ADHD, clinical trials, statistics, and data management have joined to design a double-blind sham-controlled randomized clinical trial to answer several pressing scientific and clinical questions in a way that will be credible to all. At each of 2 sites (1 university & 1 NF clinic) 70 children (total N=140) age 7 through 10 with rigorously diagnosed moderate to severe ADHD and TBR>5 will be randomized in a 3:2 ratio to active TBR downtraining by NF vs. a sham training of equal duration, intensity, and appearance. To keep both participants and study staff blind, the sham will utilize pre-recorded EEGs with the participant's artifacts superimposed. The sham will be programmed into the equipment via internet by an off-site statistician-guided person who has no contact with participants. Treatment fidelity will be trained and monitored by 2 acknowledged NF leaders in a manner that protects blinding. Multi-domain assessments at baseline, mid-treatment, treatment end, and follow-ups at 6 months, 1 year, and 2 years will include parent and teacher ratings of symptoms & impairment, neuropsychological tests,clinician ratings, and quantitative EEG as well as tests of blinding and of sham inertness. Hypotheses include that NF will improve parent- and teacher-rated inattentive symptoms (primary outcome) and other outcomes more than sham,that benefit will persist for 2 years after training, that initial TBR will moderate treatment response, and that change in TBR will mediate response. Research Domain Criteria and EEG brain changes will be explored, including relationship of TBR to clinical symptoms, executive-function impairment, and sleep.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls age 7 to 10
* IQ>80
* diagnosed DSM-5 ADHD inattentive presentation or combined presentation
* an item mean ≥1.5 sd above norms on a 0-3 metric both on parent ratings of either DSM-IV inattentive symptoms or all 18 ADHD symptoms and on teacher ratings of either inattentive symptoms or all 18 ADHD symptoms
* an eyes-open QEEG with theta-beta power ratio >4.5 at Cz or Fz

Exclusion Criteria:

* comorbid disorder requiring psychoactive medication other than FDA-approved ADHD medication
* a medical disorder requiring systemic chronic medication with confounding psychoactive effects
* sleep apnea
* restless legs syndrome
* IQ <80
* plans to move requiring school change during the next 3 months
* plans to start other ADHD treatment in the next 3 months
* antipsychotic agent in the 6 months prior to baseline assessment
* fluoxetine in the 4 weeks prior to baseline
* other psychiatric medication in the two weeks prior to baseline

  ->5 previous NF treatments
* Vitamin D deficiency will be a temporary exclusion

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L. Eugene Arnold, MD, MEd, Principal Investigator — The Ohio State University Nisonger Center; Roger deBeus, Ph.D., Principal Investigator — University of North Carolina at Asheville
Locations (2):
- United States (2):
  - University of North Carolina at Asheville, Asheville, North Carolina
  - The Ohio State University Nisonger Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ging-Jehli NR, Painter QA, Kraemer HA, Roley-Roberts ME, Panchyshyn C, deBeus R, Arnold LE. A diffusion decision model analysis of the cognitive effects of neurofeedback for ADHD. Neuropsychology. 2024 Feb;38(2):146-156. doi: 10.1037/neu0000932. Epub 2023 Nov 16. PMID 37971859
- [Derived] Ging-Jehli NR, Kraemer HC, Eugene Arnold L, Roley-Roberts ME, deBeus R. Cognitive markers for efficacy of neurofeedback for attention-deficit hyperactivity disorder - personalized medicine using computational psychiatry in a randomized clinical trial. J Clin Exp Neuropsychol. 2023 Mar;45(2):118-131. doi: 10.1080/13803395.2023.2206637. Epub 2023 May 8. PMID 37157126
- [Derived] Roley-Roberts ME, Pan X, Bergman R, Tan Y, Hendrix K, deBeus R, Kerson C, Arns M, Ging Jehli NR, Connor S, Schrader C, Arnold LE. For Which Children with ADHD is TBR Neurofeedback Effective? Comorbidity as a Moderator. Appl Psychophysiol Biofeedback. 2023 Jun;48(2):179-188. doi: 10.1007/s10484-022-09575-x. Epub 2022 Dec 16. PMID 36526924
- [Derived] Neurofeedback Collaborative Group. Neurofeedback for Attention-Deficit/Hyperactivity Disorder: 25-Month Follow-up of Double-Blind Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2023 Apr;62(4):435-446. doi: 10.1016/j.jaac.2022.07.862. Epub 2022 Dec 12. PMID 36521694
- [Derived] Neurofeedback Collaborative Group. Double-Blind Placebo-Controlled Randomized Clinical Trial of Neurofeedback for Attention-Deficit/Hyperactivity Disorder With 13-Month Follow-up. J Am Acad Child Adolesc Psychiatry. 2021 Jul;60(7):841-855. doi: 10.1016/j.jaac.2020.07.906. Epub 2020 Aug 25. PMID 32853703

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 329 children screened, 305 passed categorical and parent-rated dimensional criteria for ADHD. Of these, 235 passed the TBR screen. Of the149 completely eligible,144 were randomized, and of the 144, 2 withdrew consent for logistical reasons before any post-treatment assessment. Thus,142 subjects comprised the population for the primary analysis.
Groups:
- Neurofeedback Treatment: The intended treatment is downtraining of theta power and uptraining of beta power for 38 treatments of active NF.
  Neurofeedback treatment: Each session, the child participates in 5 training tasks. Each task lasts 5 minutes at the beginning and gradually increases to 9 minutes per task over the course of the neurofeedback as the child's attention span improves. We record four results for each of the 5 tasks:
  1. The number of half-second periods that they met the reward parameters (i.e. theta mV below threshold; beta mV above threshold)
  2. Average voltage of theta waves
  3. Average voltage of beta
  4. Average ratio of theta to beta power (TBR)
- Sham Neurofeedback Treatment: Participants assigned to sham and their trainers will be fed EEG data from pre-recorded files (recorded during live clinical NF) rather than from the participant's live signal. In order to prevent unblinding of experienced NF trainers/technicians, artifacts from the participant's EMG and EOG are blended into the pre-recorded EEG so that the trainer controlling the feedback cannot differentiate between live and simulated data. To insure trainer/technician blindness, the pre-recorded EEG will be 38 consecutive EEGs from the same age-matched clinical case so that EEGs of the sham group will also show "training progress" over successive sessions, like real NF.
  Neurofeedback treatment: Each session, the child participates in 5 training tasks. Each task lasts 5 minutes at the beginning and gradually increases to 9 minutes per task over the course of the neurofeedback as the child's attention span improves. We record four results for each of the 5 tasks.
Period: Overall Study
Arm/Group | Neurofeedback Treatment | Sham Neurofeedback Treatment
Started | 85 | 59
Completed | 84 | 58
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neurofeedback Treatment | Sham Neurofeedback Treatment | Total
Number analyzed (Participants) | 84 | 58 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.67 (1.1) | 8.51 (1.17) | 8.58 (1.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 31
  Male | 65 | 46 | 111
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 13 | 6 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 64 | 42 | 106
  Black/African American | 7 | 4 | 11
  Asian | 0 | 5 | 5
  Other | 4 | 0 | 4
  Multi-Race | 7 | 6 | 13
  Unknown | 2 | 1 | 3
Primary Living Arrangement [Count of Participants; unit: Participants]
  Parental (at least one parent) | 80 | 52 | 132
  Parental (shared custody) | 3 | 5 | 8
  Relative other than parents | 1 | 1 | 2
Number of Adults in Home [Mean (Standard Deviation); unit: average number of adults in home] | 1.94 (0.61) | 2.14 (0.78) | 2.02 (0.69)
Number of Children in Home [Mean (Standard Deviation); unit: average number of children in home] | 2.12 (1.03) | 2.12 (0.88) | 2.12 (0.97)
Primary Caregiver [Count of Participants; unit: Participants]
  Biological Mother | 67 | 49 | 116
  Biological Father | 7 | 2 | 9
  Adoptive Mother | 8 | 6 | 14
  Grandmother | 2 | 1 | 3
Child's Educational setting [Count of Participants; unit: Participants]
  Regular public school | 32 | 25 | 57
  Regular private/parochial school | 30 | 27 | 57
  Regular school + special classes | 6 | 3 | 9
  Home schooled | 3 | 0 | 3
  Charter School | 13 | 3 | 16
Child's Current grade [Count of Participants; unit: Participants]
  1 | 15 | 7 | 22
  2 | 23 | 15 | 38
  3 | 25 | 18 | 43
  4 | 12 | 13 | 25
  5 | 9 | 5 | 14
Repeated Grade [Count of Participants; unit: Participants] | 6 | 1 | 7
Number of school changes [Count of Participants; unit: Participants]
  0 | 48 | 32 | 80
  1 | 25 | 17 | 42
  2 or more | 11 | 9 | 20
Special Education Services [Number; unit: participants]
  Individual Educational Plan | 23 | 20 | 43
  504 Plan | 10 | 12 | 22
  Special accommodations | 15 | 11 | 26
ADHD Subtype [Count of Participants; unit: Participants]
  Inattentive | 31 | 20 | 51
  Combined | 53 | 38 | 91
ADHD Medication [Count of Participants; unit: Participants] | 23 | 18 | 41
Composite Conner's Subscale (Parent and Teacher) [Mean (Standard Deviation); unit: units on a scale] — The composited (averaged) scores of teacher and parent-rated subscales on the Conners-3 range from a scale of 0-3. Lower scores represent a better outcome.
  The impression indices range from 0-6. A higher score on these indices shows a measure of positive or negative bias on the parent/teacher report forms. For example, a higher score on the positive index shows a more positive bias in the ratings.
  units on a scale
    ADHD Inattentiveness | 2 (0.51) | 2.08 (0.51) | 2.03 (0.51)
    ADHD Hyperactivity-Impulsivity | 1.68 (0.77) | 1.88 (0.66) | 1.77 (0.73)
    Inattentive | 2.04 (0.52) | 2.13 (0.49) | 2.08 (0.51)
    Hyperactivity-Impulsivity | 1.71 (0.78) | 1.92 (0.64) | 1.79 (0.73)
    Learning Problems | 1.31 (0.71) | 1.18 (0.75) | 1.25 (0.73)
    Executive Functioning | 1.9 (0.62) | 1.96 (0.58) | 1.92 (0.6)
    Aggression | 0.46 (0.44) | 0.46 (0.42) | 0.46 (0.43)
    Peer Relations | 0.73 (0.67) | 0.66 (0.68) | 0.7 (0.67)
    Global Index | 1.49 (0.59) | 1.61 (0.5) | 1.54 (0.56)
    Conduct Disorder | 0.17 (0.21) | 0.15 (0.22) | 0.16 (0.22)
    Oppositional Defiant | 0.87 (0.67) | 0.92 (0.6) | 0.89 (0.64)
    Positive Impression Index | 0.32 (0.31) | 0.33 (0.32) | 0.33 (0.31)
    Negative Impression Index | 0.18 (0.23) | 0.19 (0.24) | 0.18 (0.23)
CHIPS [Number; unit: number of participants] — The Child Inventory of Psychiatric Syndomes (CHIPS) Structured diagnostic interview of child and parent
  number of participants
    Oppositional-Defiant Disorder | 41 | 30 | 71
    Specific Phobias | 15 | 9 | 24
    Generalized Anxiety Disorder | 16 | 8 | 24
    Separation Anxiety | 9 | 2 | 11
    Social Phobia | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Scores of Teacher and Parent Rated Inattentive Symptoms
Description: The primary outcome measure is the composite scores of teacher and parent-rated inattentive symptoms on the Conners-3, rated on a scale of 0-3. Lower scores represent a better outcome, with a maximum score of 3 and a minimum score of 0.
Time Frame: Assessed at Baseline, Mid-treatment (2 months), End-treatment (4 months), at 6 month follow up, at 13 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neurofeedback Treatment | Sham Neurofeedback Treatment
Number analyzed (Participants) | 84 | 58
units on a scale
  Baseline | 2.00 (0.37) | 2.08 (0.38)
  Mid-Treatment | 1.51 (0.49) | 1.60 (0.46)
  End-Treatment | 1.43 (0.51) | 1.54 (0.44)
  6 month follow up | 1.50 (0.52) | 1.52 (0.50)
  13 month follow up | 1.37 (0.56) | 1.58 (0.52)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at every visit- from baseline, at the first session of each week, and at 13-month follow up (~1.5 years).
Arm/Group | Neurofeedback Treatment | Sham Neurofeedback Treatment
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/58
Other Adverse Events (participants affected / at risk) | 75/84 | 50/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neurofeedback Treatment (N=84) | Sham Neurofeedback Treatment (N=58)
Headache (Nervous system disorders) | 9 | 5
Irritability (Social circumstances) | 7 | 7
Oppositionality (Social circumstances) | 7 | 7
Depressed mood (Psychiatric disorders) | 4 | 4
Difficulty initiating sleep (General disorders) | 6 | 2
Fatigue (General disorders) | 5 | 3
Sleep Symptoms, NOS (General disorders) | 4 | 3
Anxiety (Psychiatric disorders) | 3 | 3
Hyperactivity (Social circumstances) | 5 | 1
Aggression (Social circumstances) | 2 | 3
Agitation (General disorders) | 3 | 2
Impulsivity (Social circumstances) | 2 | 2
Crying (General disorders) | 3 | 0
Labile mood (General disorders) | 2 | 1
Sedation (Nervous system disorders) | 3 | 0
Tic disorders (Nervous system disorders) | 1 | 2
Back pain (General disorders) | 2 | 0
Behavioral, NOS (Social circumstances) | 1 | 1
Difficulty maintaining sleep (General disorders) | 1 | 1
Dizziness (General disorders) | 2 | 0
Eye pain (Eye disorders) | 2 | 0
Self-injurious behavior (General disorders) | 1 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
This study tested only one of the standard ADHD protocols, theta-beta NF. Results cannot be generalized to the other standard protocols of slow cortical potential (SCP) and sensory-motor rhythm (SMR) neurofeedback, nor fMRI neurofeedback.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT02251743/Prot_SAP_000.pdf